

Doc ID:

Revision #:1.0


| Approval | | | | |
|---|---|---|---|---|
| | Name | Position | Date | Signature |
| Revised by | Dagan Harris | VP Clinical and Regulatory affairs | 10-Feb-2024 | Noun el |
| Reviewed by | Alit Stark Inbar | VP Medical<br>Information | 10-Feb-2024 | alitStarl |
| Approved by | Alon Ironi | CEO | 10-Feb-2024 | Theranica<br>Bio-Electronics Ltd. |

Effective date of the document is from the date of approval.

| Change History | | | |
|---|---|---|---|
| Rev Rev. Date Revised by | | Revised by | Change description and reason for change |
| 1.0 | 01-Oct-2023 | Dagan Harris | Initial version |
| 2.0 | 10-Feb-2024 | Dagan Harris | Increase sample size, add additional analysis |



Doc ID:

Revision #:1.0


# **Clinical Study Protocol**

A prospective, single arm, open label post market study assessing the safety and efficacy of Nerivio for the treatment of migraine in children under the age of 12

ClinicalTrials.gov Identifier: NCT06138756

Feb 01, 2024. Rev. 2

**CONFIDENTIAL** 



Doc ID:

Revision #:1.0


## 1 TITLE PAGE

Study title: A prospective, single arm, open label post market study assessing the

safety and efficacy of Nerivio for the treatment of migraine in children

under the age of 12

Test Device: Nerivio

Indication studied: Acute treatment of migraine

Study description: Prospective, single arm, open label post market study

Sponsors: Theranica Bioelectronics Ltd

Protocol: RWE-009

Clinical Phase: Post market study

Study period: First user first treatment - May 2020

Last user last treatment - October 2023

Investigators: Dr Alit Stark Inbar

Statistician: Dr. Nira Morag-Koren.

**Koren Statistics** 

Yahadut Hadmama 6a, Herzlia Pituch, Israel



Doc ID:

Revision #:1.0


# 2 RWE-009 Study Protocol

| Title | A prospective, single arm, open label post market study assessing the safety and efficacy of Nerivio for the treatment of migraine in children under the age of 12 |
|---|---|
| Investigational Device | Nerivio is an FDA-approved remote electrical neuromodulation (REN) device for the acute and/or preventive treatment of migraine with or without aura in patients 12 years of age or older. Nerivio delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application. |
| Objectives | The study assessed the safety and efficacy of Nerivio for acute treatment of migraine in children under the age of 12. |
| Participant<br>Population | Children who were prescribed with the Nerivio device for the treatment of migraine and were under the age of 12. |
| Sample size | The sample size was defined as all Nerivio users in the Nerivio database under the age of 12 in the day of their first treatment |
| Inclusion<br>Criteria | <ul> <li>Prescribed with Nerivio device for the treatment of migraine</li> <li>Age under 12 at their first Nerivio treatment</li> <li>Treat with Nerivio at least once</li> </ul> |
| Exclusion<br>Criteria | Treatments shorter than 30 minutes |
| Study Design | A prospective, data analysis of users that met the inclusion criteria was performed. All data that were reported prior and following the treatments by the users using the electronic diary within the Nerivio application were downloaded from Theranica server in an unidentified manner. |
| Primary | Rate of Device Related Adverse Events |
| endpoint - | Incidence of device-related adverse events (DRAEs) reported by subjects. |
| Safety | <ul><li>a) Percentage of patients reporting DRAEs</li><li>b) Severity of reported DRAEs</li></ul> |



Doc ID:

Revision #:1.0


# Secondary endpoints efficacy

#### Consistent Headache Relief at 2 Hours Post-treatment.

The proportion of subjects reporting headache relief at 2 hours post-treatment in at least 50% of all their treatments.

## Consistent Freedom from Headache at 2 Hours Post-treatment.

The proportion of subjects reporting freedom from headache at 2 hours post-treatment in at least 50% of all their treatments.

## Freedom from a specific migraine associated symptom.

Freedom from a specific migraine associated symptom was calculated as the percent of patients reporting the presence of that symptom at baseline, and the lack of that symptom at 2-hours post-treatment in at least 50% of all their treatments.

Per the ICHD-3, migraine associated symptoms are:

- a) Hyper sensitivity to light (phonophobia)
- b) Hyper sensitivity to sound (phonophobia)
- c) Nausea (with or without vomiting)

## Functional disability relief

Functional disability relief was calculated as decrease of at least one level of functional disability from baseline to 2-hours post-treatment in at least 50% of all their treatments.

Disability levels are (0) none (full function), (1) mild disability, (2) moderate disability, and (3) severe disability.

## Freedom from functional disability

Freedom from functional disability was calculated as decrease from any disability level (3, 2, or 1) at baseline to no disability (i.e., return to full function) at 2-hours post-treatment in at least 50% of all their treatments.

# Exploratory efficacy endpoints

#### Use of migraine medications

Treatment patterns of Nerivio use as a standalone treatment vs. in combination with medications were extracted from the 2-hours post-treatment reports, as the percentage of treatments in which no rescue headache medications were used (Nerivio standalone), or Nerivio was used with over-the-counter (OTC) medications, or with prescription medications (Rx).

#### **Nerivio treatment stimulation intensity**

Treatment intensity (stimulation current) is set by patients via the smartphone app and automatically recorded. The average intensity over all treatments per patient was calculated to provide personal intensity levels, which was used for the analyses. Average personal intensity levels and the range for 80% of the users were calculated over the patient cohort.

## **Nerivio utilization**

Average (and/or median) of number of Nerivio treatments per month. A specific cohort of this outcome considers safety in patients who use the device at high frequency, close to the every-other-day regime of preventive treatment.



Doc ID:

Revision #:1.0


| Datasets | Intent to treat analysis set (ITT) The ITT analysis set includes all users who had at least one treatment Modified intent to treat analysis set (mITT) The mITT analysis set includes all ITT participants who had at least 2 treatments with prospective electronic diary reports at the beginning of the treatment ("baseline") and 2 hours post the beginning of the treatment. |
|---|---|
| Data Analysis | The ITT analysis set was used for the safety assessments and the mITT analysis set was used for the efficacy assessments. |

#### STATISTICAL CONSIDERATIONS FOR RWE-009 STUDY

The study hypothesis was that treatments of migraine with the Nerivio device in children will be as safe and effective as previously described in adolescents and adults.

#### DATA COLLECTION

#### **BASELINE DATA**

Baseline participant characteristics (age, gender) were collected from the Nerivio account of each participant.

#### TREATMENT DATA

Treatment data was retrieved from the Nerivio app for each treatment. Data includes automatic parameters (e.g time of treatment, location, device serial number, treatment intensity etc...) and individual information completed by the participant (pain level before and after the treatments, migraine symptoms, functional disability before and after the treatment etc...)

#### **COMPUTER SOFTWARE**

All statistical analyses and data presentations, including tabulations and listings, were performed using the SAS version 9.4 software.

## STATISTICAL ANALYSIS

## **Demographic and Baseline Analysis**

Demographic and baseline condition related characteristics will be tabulated and compared between the participant age data type. Continuous variables will be summarized by a mean, standard deviation, minimum, median and maximum and categorical variables by a count and percentage.

## **Safety Endpoints Analysis**

The rate of device related adverse event (DRAE) was calculated ad the number of reported DRAE divided by the number of participants in the study.

## **Efficacy Endpoints Analysis**

All the endpoints will be calculated for Qualified Attacks only, Qualifies treaterent was defined as

- 1 Attacks treated with Nerivio for at least 30 minutes
- 2 Pre and post treatment data wasreported by the participant for the specific treatment
- 3 No rescue medications were taken before and during the 2 hours post treatment, according to the participant report

Consistent efficacy was conducted in cases where at least two qualified treatments were performed. Patients who experienced the outcome (e.g., pain freedom) in at least 50% of their reported treatments, during which they did not report the use of rescue medications, were considered responders.

Headache pain and functional disability were rated at baseline and at 2 h post-treatment on a 4-point scale: severe, moderate, mild, or none. Migraine associated symptoms (photophobia, phonophobia, and nausea/vomiting) were marked as present or not.

Pain relief was calculated as a decrease from severe or moderate levels at baseline to mild or none at 2 h posttreatment.

Functional disability relief was calculated as any improvement in disability from baseline to 2 h posttreatment.

Pain/functional disability freedom was calculated as a decrease from any pain/disability level at baseline to none at 2 h post-treatment.

Freedom from a specific migraine-associated symptom was calculated as the percentage of patients reporting the presence of that symptom at baseline and the lack of that symptom at 2 h post-treatment. Freedom from at least one associated symptom was calculated as the percentage of patients in which one or more associated symptom(s) were reported at baseline and the lack of at least one of those symptoms at 2 h post-treatment.